CLINICAL TRIAL: NCT04382781
Title: Effect of Immunosupressive Treatment in COVID-19 Patients Whit SAM-LIKE Profile: Retrospective Cohort Study (SAM-COVID Project)
Brief Title: Immunosupressive Treatment in COVID-19 Patients
Acronym: SAM-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Spanish Network for Research in Infectious Diseases (Other)
Collaborators: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Principal Investigator, JESUS RODRIGUEZ BAÑO, Head of the Infectious Diseases Service of the HU Virgen Macarena, Spanish Network for Research in Infectious Diseases
Other Study IDs: FIS-INM-2020-03
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: COVID-19 Infection
Keywords: COVID-19; SARS-CoV-2; Immunosuppressive; Immunoglubulins
MeSH Terms: conditions — COVID-19 | interventions — Immunosuppressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- COVID-19 infection: Consecutive patients admitted to Spanish hospitals with laboratory-confirmed COVID-19 infection by real-time polymerase chain reaction (RT-PCR) assay for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) who showed clinical and analytical data suggestive of macrophage activation syndrome during admission until March 30, 2020 .
  Interventions: Drug: NO-Immunosuppressive; Drug: Immunosuppressive; Drug: Immunoglubulins

INTERVENTIONS:
Drug: NO-Immunosuppressive — Patients not receiving immunosuppressive drugs
Drug: Immunosuppressive — Patients receiving immunosuppressive drugs (overall, and specific drugs)
Drug: Immunoglubulins — Patients receiving immunoglubulins

SUMMARY:
SAM-COVID is a retrospective cohort study that aims to determine the impact of immunosuppressive drugs and immunoglubulins in the outcome of patients with COVID-19.

DETAILED DESCRIPTION:
SAM-COVID is a retrospective cohort study of patients admitted to 66 Spanish hospitals with laboratory-confirmed COVID-19 infection by real-time polymerase chain reaction (RT-PCR) assay for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) presenting during admission with clinical and laboratory data suggestive of macrophage activation syndrome with the objective to investigate whether the use of immunosuppressive drugs (including high-dose steroids, tocilizumab, sarilumab, anakimra) or immunoglobulins in avoiding the need for invasive mechanical ventilation or in-hospital death.

The Ethics Committee for Research of Virgen Macarena and Virgen del Rocío University Hospitals approved the study and waived the need to obtain informed consent.

The data source was the electronic medical records. All data were entered directly by personnel at each institution using an online case report form (CRF), that satisfied local requirements of data confidentiality.

The variables registered included administrative data, epidemiological information, type of clinical specimen in which the diagnosis was confirmed, demographics, comorbidities and current medications, signs and symptoms at admission, baseline laboratory tests results and at day 0, chest X-ray findings at baseline and during follow-up, medications with potential activity against COVID-19, supportive treatments including oxygen therapy, use of immunosuppressant medications or immunoglobulins, and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) admitted because of COVID-19 confirmed by PCR in nasopharyngeal swab or lower respiratory tract sample and presenting on a specific date (day 0) one clinical and one laboratory criteria of the following:

Clinical criteria:

* Temperature ≥38ºC.
* Worsening in oxygen requirements to achieve O2 saturation >92%.

Laboratory criteria:

* Ferritin >2000 ng/mL or increment in >1000 ng/ML since admission.
* D-dimer >1500 µg/mL (or duplicate in 24h)
* IL6 >50 pg/mL.

Exclusion Criteria:

* Mechanical ventilation in day 0.
* Decision of provide only palliative care before day 0.
* Use of systemic steroids, tocilizumab, other immunosupressors, or immunoglobulins before day 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to Spanish hospitals with laboratory-confirmed COVID-19 infection by real-time polymerase chain reaction (RT-PCR) assay for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) who showed clinical and analytical data suggestive of macrophage activation syndrome during admission until March 30, 2020 .
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Invasive ventilation or death | Up to 21 days
  Days until invasive mechanical ventilation or death, whatever happened first.

SECONDARY OUTCOMES:
Ventilation | Up to 21 days
  Days until mechanical ventilation
Death | Up to 21 days
  Days until death
Secondary infections | Up to 21 days
  Proportion of patients developing secondary infections
Digestive tract hemorrhage | Up to 21 days
  Proportion of patients with digestive tract hemorrhage
Change in 7 points scale | Day 21
  Proportion of patients with imnprovement in 2 or more points in 7-point scale by WHO

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Virgen Macarena, Seville, Spain

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT04382781/Prot_SAP_000.pdf